CLINICAL TRIAL: NCT05549505
Title: An Open-label, Randomized, Non-comparative Phase 2 Study of ARV-471 or Anastrozole in Post-menopausal Women With ER+/HER2- Breast Cancer in the Neoadjuvant Setting
Brief Title: A Trial Using ARV-471 or Anastrozole in Post-Menopausal Women With Breast Cancer Prior to Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arvinas Inc. (Industry)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARV-471-BC-201; C4891025 (Other: Pfizer)
Record Dates: First submitted 2022-09-07; First posted 2022-09-22 (Actual); Results first posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer
Keywords: Early breast cancer; Localized breast cancer; Untreated breast cancer; Pre-operative breast cancer; Treatment-naïve breast cancer; Neoadjuvant; Estrogen receptor; Estrogen receptor positive; ER+; Hormone positive; Hormone receptor positive; HR+; human epidermal growth factor receptor 2 negative; HER2-; ARV-471; Anastrozole; Arimidex; Aromatase inhibitor; Vepdegestrant; PF-07850327
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: ARV-471 (Experimental) (Experimental): Participants received 200 mg ARV-471 (2*100 mg tablets) once daily for approximately 5.5 months prior to undergoing surgical resection (no later than Cycle 6 Day 18 [C6D18] + 14 days).
  Interventions: Drug: ARV-471; Procedure: Surgical resection of breast tumor
- Arm B: Anastrozole (Active Comparator): Participants received 1 mg Anastrozole tablet orally once daily for approximately 5.5 months prior to undergoing surgical resection (no later than C6D18 + 14 days).
  Interventions: Drug: Anastrozole; Procedure: Surgical resection of breast tumor

INTERVENTIONS:
Drug: ARV-471 — 100 mg tablet
  Other Names: Vepdegestrant; PF-07850327
  Arms: Arm A: ARV-471 (Experimental)
Drug: Anastrozole — 1 mg tablet
  Other Names: Arimidex
  Arms: Arm B: Anastrozole
Procedure: Surgical resection of breast tumor — Surgical resection approximately 5.5 months after starting treatment (C6D18 ± 14 days)

SUMMARY:
This trial is a Phase 2 neoadjuvant study evaluating ARV-471 or anastrozole in post-menopausal women with estrogen receptor positive/ human epidermal growth factor receptor 2 (ER+/HER2)- localized breast cancer.

DETAILED DESCRIPTION:
This is a Phase 2, open-label, randomized, non-comparative proof of concept study of ARV-471 or anastrozole in participants with ER+/HER2- breast cancer amenable to definitive surgical resection. The main goal of this study is to evaluate the biological activity of ARV-471 and anastrozole, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal females ≥ 18 years.
* Histologically or cytologically confirmed ER+ and HER2- breast cancer (per local assessment). ER and HER2 status must be documented:

  * ER+ disease, with ER staining of ≥ 10% of tumor cell nuclei by immunohistochemistry (IHC) per American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) guidelines.
  * HER2- disease by either IHC or in situ hybridization per ASCO/CAP guidelines.
  * Ki-67 score ≥ 5%, analyzed locally.
* Clinical T1c-T4c, N0-N2, M0 breast cancer amenable to definitive surgical resection, without bilateral breast ductal carcinoma in situ or invasive breast cancer.
* The primary tumor must be at least 1.5 cm by imaging.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Willingness to undergo a screening biopsy, an on-treatment biopsy and surgical resection.

Exclusion Criteria:

* Any other active malignancy within 3 years prior to enrollment, except for adequately treated basal cell or squamous cell skin cancer, or cervical carcinoma in situ.
* Any of the following in the previous 6 months: Myocardial infarction; Severe unstable angina; Coronary/peripheral artery bypass graft; Symptomatic congestive heart failure (New York Heart Association class III or IV); Cerebrovascular accident; Transient ischemic attack; Symptomatic pulmonary embolism or other clinically significant episode of thromboembolism.
* Any of the following in the previous 6 months: Congenital long QT syndrome; Torsade de Pointes; Sustained ventricular tachyarrhythmia and ventricular fibrillation; Left anterior hemiblock (bifascicular block); Ongoing cardiac dysrhythmias of NCI CTCAE ≥ Grade 2; Atrial fibrillation of any grade (≥ Grade 2 in the case of asymptomatic lone atrial fibrillation).
* corrected QT (Fridericia method) (QTcF) > 470 msec.
* Active, uncontrolled bacterial, fungal or viral infection, including (but not limited to) hepatitis B virus (HBV), hepatitis C virus (HCV), and known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
* Active inflammatory gastrointestinal disease, chronic diarrhea, known uncontrolled diverticular disease, or previous gastric resection or lap band surgery.
* Cirrhosis meeting criteria for Child Pugh B and C.
* Prior treatment for breast cancer including systemic therapy (eg, chemotherapy, hormonal therapy), radiation, surgery, or any investigational agents.
* Any live vaccines within 14 days of planned start of first dose of study drug.
* Major surgery (as defined by the Investigator) within four weeks of first dose of study drug.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-07-13 (Actual); Study Completion 2024-07-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (39):
- United States (13):
  - Clinical Trial Site, Springdale, Arkansas
  - Clinical Trial Site, Los Angeles, California
  - Clinical Trial Site, Torrance, California
  - Clinical Trial Site, Van Nuys, California
  - Clinical Trial Site, Fort Lauderdale, Florida
  - Clinical Trial Site, Fort Myers, Florida
  - Clinical Trial Site, Orlando, Florida
  - Clinical Trial Site, West Palm Beach, Florida
  - Clinical Trial Site, Iowa City, Iowa
  - Clinical Trial Site, Springfield, Massachusetts
  - Clinical Trial Site, St Louis, Missouri
  - Clinical Trial Site, Nashville, Tennessee
  - Clinical Trial Site, Tacoma, Washington
- Georgia (2):
  - Clinical Trial Site, Batumi
  - Clinical Trial Site, Tbilisi
- Germany (11):
  - Clinical Trial Site, Augsburg
  - Clinical Trial Site, Berlin
  - Clinical Trial Site, Bonn
  - Clinical Trial Site, Bottrop
  - Clinical Trial Site, Chemnitz
  - Clinical Trial Site, Dresden
  - Clinical Trial Site, Erlangen
  - Clinical Trial Site, Essen
  - Clinical Trial Site, Esslingen am Neckar
  - Clinical Trial Site, Mannheim
  - Clinical Trial Site, Paderborn
- Spain (13):
  - Clinical Trial Site, A Coruña, Galicia
  - Clinical Trial Site, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Clinical Trial Site, Alicante
  - Clinical Trial Site, Barcelona
  - Clinical Trial Site, Castelló
  - Clinical Trial Site, Córdoba
  - Clinical Trial Site, Granada
  - Clinical Trial Site, Lleida
  - Clinical Trial Site, Madrid
  - Clinical Trial Site, Manresa
  - Clinical Trial Site, Seville
  - Clinical Trial Site, Valencia
  - Clinical Trial Site, Zaragoza

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 152 participants were enrolled.
Period: Overall Study
Arm/Group | Arm A: ARV-471 (Experimental) | Arm B: Anastrozole
Started | 102 | 50
Treated | 101 | 48
Completed | 94 | 41
Not Completed | 8 | 9
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Other: Miscellaneous | 3 | 6

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all the enrolled participants who were randomized.
Groups:
- Arm A: ARV-471 (Experimental): Participants received 200 mg ARV-471 (2*100 mg tablets) once daily for approximately 5.5 months prior to undergoing surgical resection (no later than C6D18 + 14 days).
- Total: Total of all reporting groups
Arm/Group | Arm A: ARV-471 (Experimental) | Arm B: Anastrozole | Total
Number analyzed (Participants) | 102 | 50 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (9.23) | 66.8 (8.31) | 67.2 (8.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102 | 50 | 152
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 38 | 23 | 61
  Not Hispanic or Latino | 59 | 25 | 84
  Unknown or Not Reported | 5 | 2 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 98 | 46 | 144
  Other | 0 | 1 | 1
  Unknown or Not Reported | 2 | 0 | 2
Percentage of Tumor Cells Positive for Ki -67 [Mean (Standard Deviation); unit: Percentage of tumor cells with Ki67] — Ki-67 expression assessed by immunohistochemical staining in a central laboratory. Population: Only participants with evaluable central Ki-67 results included in the analysis.
  Percentage of tumor cells with Ki67
    number analyzed (Participants) | 100 | 48 | 148
    (all) | 20.6 (14.01) | 20.1 (12.25) | 20.4 (13.42)

OUTCOME MEASURES:

1. Primary Outcome: Percent Reduction in Ki-67 Expression From Baseline to Day 15 in Tumor Biopsies
Description: Tumor biopsy Ki-67 expression (% of tumor cells that are positive for Ki-67) at baseline and Cycle 1 Day 15 (C1D15) was collected. Ki-67 expression was assessed by immunohistochemical staining in a central laboratory. The log-transformed Ki-67 after approximately 2 weeks of treatment as a percentage of the baseline value, ie, the ratio between the Ki-67 measurements obtained from C1D15 visit and baseline was modelled using a generalized linear model (GLM) with both stratification factors (ie, baseline Ki-67 score and the tumor size) and treatment as co-variates. The treatment effects were back transformed into geometric means and their Confidence Intervals. The percent change, in other words, relative reduction, of Ki-67 after 2 weeks of treatment is reported as the complement of the ratio between the Ki-67 measurement from C1D15 and baseline, that is 100% × (1 - geometric mean ratio between Ki-67 at C1D15 and Ki-67 at baseline).
Time Frame: Baseline (during screening, prior to Day 1) and Day 15
Population: Ki-67 Evaluable Set included all enrolled participants who were randomized and received at least one dose of study treatment and had evaluable central Ki-67 measurements other than '0' or '< 1' from baseline and evaluable Ki-67 measurements from C1D15 visits.
Measure: Number (95% Confidence Interval); unit: Percent reduction
Arm/Group | Arm A: ARV-471 (Experimental) | Arm B: Anastrozole
Number analyzed (Participants) | 93 | 46
Percent reduction | 71.4 [60.6 to 79.3] | 72.9 [57.8 to 82.6]

2. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs and TEAEs Leading to Study Drug Discontinuation
Description: An AE is any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study intervention. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. A TEAE is an AE that emerges or worsens on/after the first dose of ARV-471/Anastrozole to 30 days after the last administration of the study intervention (ie, study drug treatment or surgical resection, whichever occurs last).
Time Frame: From signing of consent to minimum of 30 days after last administration of study drug (up to approximately 6.5 months)
Population: Safety Analysis Set which consisted of all enrolled participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: ARV-471 (Experimental) | Arm B: Anastrozole
Number analyzed (Participants) | 101 | 48
Participants
  TEAEs | 82 | 37
  Serious TEAEs | 4 | 5
  TEAEs leading to study drug discontinuation | 3 | 4

3. Secondary Outcome: Pathologic Stage at the Time of Surgical Resection
Description: Local pathological assessment of the tissue from surgical resection (performed after approximately 5.5 months of treatment), at minimum, included pathologic stage (ypT and ypN stage) as described in the Laboratory Manual. Participants were analysed based on the current American Joint Committee on Cancer (AJCC) staging system as follows:
  * Pathologic Tumor - post-neoadjuvant therapy pathologic tumor categorization (ypT): (ypTx, ypT0, ypTis, ypT1mi, ypT1a, ypT1b, ypT1c, ypT2, ypT3, ypT4a, ypT4b, ypT4c).
  * Pathological Lymph Nodes - post-neoadjuvant therapy pathologic node categorization (ypN): (ypNX, ypN0, ypN0(i+), ypN0(mol+), ypN1, ypN1mi, ypN1a, ypN1b, ypN1c, ypN2, ypN2a, ypN2b, ypN3, ypN3a, ypN3b, ypN3c).
  * ypT0 / ypN0 indicates no evidence of disease and the progressive grades indicate increasing size of tumor and increasing area of lymph node involvement respectively and ypTx/ypNX indicates non-measurable disease.
Time Frame: At Cycle 6 Day 18 (approximately 5.5 months), each cycle is 28 days
Population: Full Analysis Set included all the enrolled participants who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: ARV-471 (Experimental) | Arm B: Anastrozole
Number analyzed (Participants) | 102 | 50
Participants
  Pathologic Tumor ypTx | 0 | 0
  Pathologic Tumor ypT0 | 1 | 0
  Pathologic Tumor ypTis | 1 | 0
  Pathologic Tumor ypT1mi | 1 | 0
  Pathologic Tumor ypT1a | 6 | 1
  Pathologic Tumor ypT1b | 7 | 2
  Pathologic Tumor ypT1c | 36 | 14
  Pathologic Tumor ypT2 | 33 | 21
  Pathologic Tumor ypT3 | 4 | 2
  Pathologic Tumor ypT4a | 1 | 0
  Pathologic Tumor ypT4b | 0 | 0
  Pathologic Tumor ypT4c | 0 | 0
  Pathologic Tumor Not Evaluable | 12 | 10
  Pathological Lymph Nodes ypNX | 0 | 0
  Pathological Lymph Nodes ypN0 | 51 | 20
  Pathological Lymph Nodes ypN0(i+) | 0 | 0
  Pathological Lymph Nodes ypN1 | 5 | 4
  Pathological Lymph Nodes ypN0(mol+) | 0 | 0
  Pathological Lymph Nodes ypN1mi | 4 | 3
  Pathological Lymph Nodes ypN1a | 21 | 6
  Pathological Lymph Nodes ypN1b | 0 | 0
  Pathological Lymph Nodes ypN1c | 1 | 0
  Pathological Lymph Nodes ypN2 | 2 | 2
  Pathological Lymph Nodes ypN2a | 3 | 4
  Pathological Lymph Nodes ypN2b | 0 | 0
  Pathological Lymph Nodes ypN3 | 0 | 0
  Pathological Lymph Nodes ypN3a | 3 | 1
  Pathological Lymph Nodes ypN3b | 0 | 0
  Pathological Lymph Nodes ypN3c | 0 | 0
  Pathological Lymph Nodes Not evaluable | 12 | 10

4. Secondary Outcome: Pathological Complete Response(pCR) Rate at the Time of Surgical Resection
Description: pCR is defined as no invasive cancer in the breast and sampled axillary lymph nodes following completion of neoadjuvant systemic therapy (ie, Pathologic Tumor - ypT = ypT0 or ypTis, and Pathologic Lymph Nodes - ypN = ypN0 in the current American Joint Committee on Cancer (AJCC) staging system). pCR rate is the percentage of participants with pCR.
Time Frame: At Cycle 6 Day 18 (approximately 5.5 months), each cycle is 28 days
Population: Full Analysis set included all the enrolled participants who were randomized.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: ARV-471 (Experimental) | Arm B: Anastrozole
Number analyzed (Participants) | 102 | 50
percentage of participants | 1 | 0

5. Secondary Outcome: Number of Participants With Modified Preoperative Endocrine Prognostic Index (mPEPI) Score of 0 at the Time of Surgical Resection
Description: Modified Pre-operative Endocrine Prognostic Index (mPEPI) score is an investigational prognostic tool used to predict the risk of breast cancer recurrence. It will be derived from factors assigned a numerical score following Neoadjuvant endocrine treatment (NET). The factors include pathologic tumor size, and lymph node status and Ki67 expression in the surgical specimen. Total mPEPI score (mPEPI_T) per participant is the sum of mPEPI score of each factor.
  mPEPI score of 0 indicates Pathological tumor size T1-T2, no lymph nodes and Ki67 level of 0%-2.7%, 1 indicates: Ki67 level >2.7%-7.3%, 2 indicates Ki67 level >19.7%-53.1% and 3 indicates: tumor sizeT3-T4, presence of lymph nodes and Ki67 level >53.1%.
Time Frame: At Cycle 6 Day 18 (approximately 5.5 months), each cycle is 28 days
Population: Full Analysis Set included all the enrolled participants who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: ARV-471 (Experimental) | Arm B: Anastrozole
Number analyzed (Participants) | 102 | 50
Participants | 21 | 10

6. Secondary Outcome: Breast Conserving Surgery (BCS) Rate
Description: Breast conserving surgery (BCS) Rate is the percentage of participants received breast conserving surgery.
Time Frame: At Cycle 6 (from Day 141 to Day 168), each cycle is 28 days
Population: Full Analysis Set included all the enrolled participants who were randomized.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Arm A: ARV-471 (Experimental) | Arm B: Anastrozole
Number analyzed (Participants) | 102 | 50
Percentage of participants | 69.6 [60.1 to 77.7] | 54.0 [40.4 to 67.0]

7. Secondary Outcome: Radiographic Response Per Modified Response Evaluation Criteria in Solid Tumors (mRECIST) in Primary Tumor During Cycle 6
Description: The number of participants with Complete Response (CR), Partial Response (PR), Stable Disease (SD), Progressive Disease (PD), Not Evaluable (NE) per mRECIST calculated. CR = disappearance of all target lesions, PR is >=30% decrease in sum of diameters of target lesions, progressive disease (PD) is >=20% increase in sum of diameters of target lesions, stable disease (SD) is <30% decrease or <20% increase in sum of diameters of target lesions.
Time Frame: At Cycle 6 (from Day 141 to Day 168), each cycle is 28 days
Population: Full Analysis Set included all the enrolled participants who were randomized.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: ARV-471 (Experimental) | Arm B: Anastrozole
Number analyzed (Participants) | 102 | 50
Participants
  CR | 5 | 4
  PR | 37 | 17
  Stable Disease | 38 | 16
  Progressive disease | 3 | 1
  NE | 19 | 12

8. Secondary Outcome: Percentage Change From Baseline at Cycle 6 Day 1 in Caliper Measurement of the Primary Tumor
Description: The percentage change from the baseline of the primary breast tumor size in physical exam calculated in caliper measurement. Caliper-based response is the maximum percentage decrease or minimum percentage increase if there is no decrease per participant.
Time Frame: Baseline (Day 1) and Cycle 6 Day 1 (At Day 141), each cycle is 28 days
Population: Full Analysis Set included all the enrolled participants who were randomized. Here "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Arm A: ARV-471 (Experimental) | Arm B: Anastrozole
Number analyzed (Participants) | 45 | 19
Percent change | -32.35 (23.739) | -42.88 (18.041)

ADVERSE EVENTS:
Time Frame: Adverse Events: From first study drug administration up to approximately 6.5 months. All-cause mortality: From randomization up to approximately 6.5 months.
Description: Adverse events were collected for the Safety Analysis Set consisting of all enrolled participants who received at least 1 dose of study intervention. For All-Cause Mortality, events were collected from the Full Analysis Set, which included all the enrolled participants who were randomized.
Arm/Group | Arm A: ARV-471 (Experimental) | Arm B: Anastrozole
All-Cause Mortality (participants affected / at risk) | 0/102 | 0/50
Serious Adverse Events (participants affected / at risk) | 4/101 | 5/48
Other Adverse Events (participants affected / at risk) | 72/101 | 32/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: ARV-471 (Experimental) (N=101) | Arm B: Anastrozole (N=48)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Mental status change (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: ARV-471 (Experimental) (N=101) | Arm B: Anastrozole (N=48)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 7 (7) | 2 (2)
Constipation (Gastrointestinal disorders) | 16 (19) | 3 (3)
Nausea (Gastrointestinal disorders) | 15 (16) | 1 (2)
Asthenia (General disorders) | 21 (24) | 5 (5)
Fatigue (General disorders) | 13 (14) | 3 (3)
COVID-19 (Infections and infestations) | 6 (6) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4) | 3 (3)
Urinary tract infection (Infections and infestations) | 8 (10) | 1 (1)
Alanine aminotransferase increased (Investigations) | 6 (6) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 8 (10) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (16) | 15 (15)
Dizziness (Nervous system disorders) | 5 (5) | 3 (3)
Headache (Nervous system disorders) | 8 (10) | 1 (1)
Insomnia (Psychiatric disorders) | 9 (10) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Hot flush (Vascular disorders) | 25 (28) | 10 (10)
Hypertension (Vascular disorders) | 12 (18) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-01-09): https://cdn.clinicaltrials.gov/large-docs/05/NCT05549505/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT05549505/SAP_001.pdf